CLINICAL TRIAL: NCT03111563
Title: Effectiveness of Warm Saline Distension Media on Relieving Pain in Office Hysteroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Melad Eskander, Sohag, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WSDM
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Hysteroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- warm saline (Other): case group ,
  Interventions: Other: Warm saline distension media in office hysteroscopy
- room temperature (Other): control group
  Interventions: Other: Warm saline distension media in office hysteroscopy

INTERVENTIONS:
Other: Warm saline distension media in office hysteroscopy — warm saline distension media in office hysteroscopy

SUMMARY:
The aim of the study is to compare the effectiveness of warm saline distension media versus room temperature saline distension media on relieving pain in office hysteroscopy .

DETAILED DESCRIPTION:
Research hypothesis :

In women undergoing diagnostic hysteroscopy, warm saline distension media may be effective in decreasing the pain during the procedure .

Research question :

In women undergoing diagnostic hysteroscopy, does warm saline distension media decrease the pain during the procedure ?

Aim of the work :

- This study aim to assess the efficacy of warm saline distension media in decreasing the pain in women undergoing diagnostic hysteroscopy

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-40 years old (premenopausal women ).
2. Normal cervical morphology during speculum examination.
3. Women complaining of abnormal uterine bleeding
4. Women underging the procedure to evaluate the endocervical canal, uterine cavity and tubal ostia because of infertility.
5. Suspected mullerian anomalies.

Exclusion Criteria:

* a. Pregnancy. b. Suspected acute pelvic inflammatory disease. c. Past history of medical disorders, especially associated with neuropathies, e.g. diabetes, chronic kidney disease, etc.

  d. History of vaginal pruritis, discharge, dysuria, dysmenorrhea, dyspareunia or chronic pelvic pain.

  e. Presence of pain, profuse bleeding or other symptoms at the time of the procedure.

  f. History of uterine surgery that occurred less than 1 month previously. g. History of previous cervical procedures. h. Administration of general, cervical or paracervical anesthesia. i. Administration of sedatives. j. Any use of analgesic agents before the procedure. k. Cervical preparation by misoprostol before procedure orally or vaginally for cervical ripening to improve the likelihood of successful cervical dilation and decrease intraoperative pain .

  l. Need for cervical dilatation during procedure. m. Need for biopsy or any operative intervention during the procedure.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
assesment of pain immediately at the end of the procedure and 15 minutes after it | immediately after the procedure and 15 minutes after the end of it
  d. The degree of pain that the patient feels in the procedure will be estimated by using visual analoge scale (VAS) (figure 1) at 2 times: At the end of the procedure and at 15 minutes after the examination. The patient makes a mark on the VAS line to indicate the intensity of her pain. The distance from the zero point to the marked point is measured using a graduated ruler. Each pain assessment is made on a separate line.

SECONDARY OUTCOMES:
patient satisfaction | during procedure
  Patients' satisfaction will be evaluated as the percentage of patients who would undergo the examination again using the same method
time taken to complete the procedure | during procedure
  The time taken to perform the examination is measured in minutes, from introduction from the cervix.of the hysteroscope into the vagina until removing it

IPD SHARING:
Plan to Share IPD: No